CLINICAL TRIAL: NCT06595719
Title: Assessing Gut Microbiota, Mucosal Healing Markers, and Metabolites in Mild to Moderate Ulcerative Colitis Treated With Multi-Strain Probiotics
Brief Title: Multi-Strain Probiotics Supplementation With Standard Care in Mild to Moderate Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2023-852
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
Keywords: Probiotics; Inflammatory Bowel Disease; Gut microbiota
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics with standard care (Experimental): 62 mild to moderate UC patients were supplemented with multi-strain probiotics consisting of 6 active strains from Bifidobacterium and Lactobacillus species for 12 weeks.
  Interventions: Dietary Supplement: Multi-Strain Probiotics
- Placebo with standard care (Placebo Comparator): 62 mild to moderate UC patients were supplemented with placebo, containing no active bacteria strains for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-Strain Probiotics — Each sachet of the multi-strain probiotics contain 30 billion CFU of 6 strains which includes Lactobacillus acidophilus BCMC®12130, Lactobacillus casei subsp BCMC®12313, Lactobacillus lactis BCMC®12451, Bifidobacterium bifidum BCMC®02290, Bifidobacterium infantis BCMC®02129, Bifidobacterium longum BCMC®02120
  Arms: Probiotics with standard care
Dietary Supplement: Placebo — Replicate for multi-strain probiotics without any active ingredients
  Arms: Placebo with standard care

SUMMARY:
Probiotics are one of the adjunctive treatments that have been extensively explored for Ulcerative colitis (UC) disease management. Probiotics, a group of beneficial bacteria, can bring various health benefits when adequately supplied to the body, especially for gut wellness. In particular, for UC patients, gut dysbiosis is one of the contributing factors in their pathogenesis. Thus, the supplementation of probiotics in combination with standard treatment can potentially help in relieving symptoms as well as promoting mucosal healing for long-term remission.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) has progressively risen globally, becoming more prevalent in recent years. Crohn's disease (CD) and UC are classified as two of IBD variations resulting in range of symptoms that can negatively impact patients' quality of life. The underlying cause of UC is complicated, encompassing genetic, environmental, and immunological factors. Despite breakthroughs in medical treatment, obtaining and maintaining remission in UC remains a substantial challenge, especially for people with mild to moderate disease severity. Standard treatment for UC consists of anti-inflammatory drugs, antibiotics, immunosuppressants, and, in severe instances, biologic therapy and possibly surgery. While these procedures have proven effective, a significant proportion of patients endure ongoing symptoms or undesirable consequences, emphasizing the need for alternative or supplementary therapeutic options.

In recent years, studies have focused on the gut microbiota as an important contributor in the pathophysiology of UC. Individuals with UC frequently exhibit altered microbial composition and dysbiosis, implying a possible role for gut microbiome-modulating therapies. Probiotics, which are live microorganisms that provide health advantages have emerged as a viable area for research in UC management. The rationale for using probiotics in UC lies in their potential to restore microbial balance, strengthen the intestinal barrier, and modulate the immune response. Previous studies have shown varying degrees of success with probiotics administration in terms of clinical and laboratory outcomes.

This proposed research seeks to contribute to the growing body of knowledge on the role of probiotics in UC by evaluating the efficacy of a multi-strain probiotic supplement. By combining these probiotics with standard care, we aim to explore the synergistic effects that may lead to improved clinical outcomes, endoscopic remission, and enhanced quality of life in individuals with mild to moderate UC. Understanding the impact of multi-strain probiotics on UC could provide clinicians with a valuable adjunctive tool for UC treatment strategies. Furthermore, elucidating the underlying mechanisms by which probiotics exert their effects enable better knowledge regarding the interplay between the gut microbiota and UC management. Thus, it can bring benefits to both patients and health institutions which helped in reducing the cost and maintaining long term remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC established by previous colonoscopy, with consistent histology, and clinical course.
* UC involving at least the rectosigmoid, actively confirmed by colonoscopy at the beginning of the study.
* Mild to moderate disease activity, defined as a PMS ranging from 3-8.
* Use of medication at least 4 weeks prior to study.

Exclusion Criteria:

* Crohn's disease or pouchitis.
* Severe disease activity as defined in PMS, more than 8.
* Use of antibiotics within the last 2 weeks before study entry.
* Change in dose of medication within the last 4 weeks before study entry and throughout the 12-week study period.
* Use of probiotics preparation either prescribed or over the counter within 2 weeks before the study entry.
* Use of NSAIDs for 1 week before and throughout the 12-week study period.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome analysis | 12 weeks
  The composition, diversity, and core microbiome of the gut bacterial community were identified via 16S rRNA sequencing and compared before and after taking multi-strain probiotics or placebo.
Faecal Calprotectin Level | 12 weeks
  Level of faecal calprotectin (mg/kg) measured before and after treatment with multi-strain probiotics or placebo, indicating levels of intestinal inflammation.
C-reactive Protein (CRP) Level | 12 weeks
  Level of CRP (mg/dl) measured before and after treatment with multi-strain probiotics or placebo, reflecting changes in systemic inflammation.
Erythrocyte Sedimentation Rate (ESR) Level | 12 weeks
  Rate of erythrocyte sedimentation (mm/hr) measured before and after treatment with multi-strain probiotics or placebo, as a marker of inflammation.
Change in White Blood Cell (WBC) Count | 12 weeks
  Number of participants with changes in WBC count (x10^9/L) measured before and after treatment with multi-strain probiotics or placebo, to assess immune response and inflammation levels.
Change in Serum Metabolite Profile | 12 weeks
  Identification and quantification of serum metabolites via Liquid Chromatography-Mass Spectrometry (LC-MS) before and after treatment with multi-strain probiotics or placebo. The changes in metabolite concentrations will be compared to assess the metabolic response to the intervention.
Change in Proinflammatory Cytokine Gene Expression | 12 weeks
  Quantification of IL5, IL6, IL13, IL33, and TNFα gene expression using quantitative PCR (qPCR) before and after treatment with multi-strain probiotics or placebo. The changes in gene expression levels will be compared to evaluate the impact on proinflammatory cytokines.

SECONDARY OUTCOMES:
Partial Mayo score (PMS) | 12 weeks
  Assessment of disease severity using the Partial Mayo Score, a scale ranging from 0 to 9, where higher scores indicate worse disease severity. The PMS was used during the screening process to identify mild to moderate UC patients, and was also measured after 12 weeks of intervention during post-treatment sample collection to evaluate changes in disease severity.
International Physical Activity Questionnaire (IPAQ) | 12 weeks
  Physical activity was assessed using the International Physical Activity Questionnaire (IPAQ), completed by participants before and after treatment with multi-strain probiotics or placebo. The total weekly minutes for each domain (e.g., walking, moderate activity, vigorous activity) will be summed to estimate the participant's overall physical activity level.
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | 12 weeks
  Quality of Life (QoL) was assessed through patient-completed questionnaires before and after treatment with multi-strain probiotics or placebo. Total scores will be calculated, with higher or lower scores indicating the patient's overall QoL. The change in scores will be used to determine the impact of the intervention on QoL.
Three Days Food Record | 12 weeks
  Dietary intake over the past three days was recorded by participants using a Three-Days Food Record before and after treatment with multi-strain probiotics or placebo. The data will be used to assess changes in participants' dietary patterns and nutrient intake prior to sample collection.
Diet History Questionnaire | 12 weeks
  At the end of the 12-week intervention, participants completed a Diet History Questionnaire to report their intake of probiotics-based foods, including conventional and local foods. This data will provide insight into the participants' consumption of probiotics-based foods during the intervention period, helping to account for potential bias in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
No The investigators are bound to the Institutional Review Board Universiti Kebangsaan Malaysia Medical Research Ethics Committee rules and regulations where recruited patients identity and data are kept confidential and will only be allowed to access by the research team.